CLINICAL TRIAL: NCT07378423
Title: Questionnaire on Congenital Cancer Signs Through Self-Assessment (QUOCCAS)
Brief Title: Questionnaire on Congenital Cancer Signs Through Self-Assessment
Acronym: QUOCCAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Berner Stiftung für krebskranke Kinder und Jugendliche (Unknown); Fondation CANSEARCH (Unknown); Childhood Cancer Switzerland (Unknown); Zoé4Life (Unknown); Swiss Cancer League (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2025-01346
Record Dates: First submitted 2025-11-18; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cancer Predisposition Syndromes; Pediatric Cancer; Childhood Neoplasms; Hereditary Cancer Syndromes
Keywords: Cancer Predisposition Syndrome (CPS); Pediatric Oncology; Childhood Cancer; Genetic Testing; Whole-Exome Sequencing (WES); Screening Tool; Patient-Reported Outcomes; Genetic Literacy; Whole-Genome Sequencing (WGS)
MeSH Terms: conditions — Neoplasms; Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Visit Preparation (PVP) Brochure + QUOCCAS Questionnaire (Experimental): Participants will receive the educational Pre-Visit Preparation (PVP) brochure before completing the QUOCCAS questionnaire. They will also provide a saliva or blood sample for germline genetic sequencing and complete follow-up surveys.
  Interventions: Behavioral: Pre-Visit Preparation (PVP) Brochure; Diagnostic Test: QUOCCAS Questionnaire; Diagnostic Test: Germline genetic sequencing for Cancer Predisposition Syndromes (CPS); Diagnostic Test: MIPOGG Assessment
- QUOCCAS Questionnaire Only (Active Comparator): Participants will complete the QUOCCAS questionnaire without receiving the Pre-Visit Preparation (PVP) brochure. They will also provide a saliva or blood sample for germline genetic sequencing and complete follow-up surveys.
  Interventions: Diagnostic Test: QUOCCAS Questionnaire; Diagnostic Test: Germline genetic sequencing for Cancer Predisposition Syndromes (CPS); Diagnostic Test: MIPOGG Assessment

INTERVENTIONS:
Behavioral: Pre-Visit Preparation (PVP) Brochure — Participants receive a Pre-Visit Preparation (PVP) brochure containing information about cancer predisposition syndromes, genetic testing, and implications for care. The brochure is provided before completion of the QUOCCAS questionnaire and is designed to improve caregiver knowledge, engagement, and satisfaction with care.
  Other Names: Educational Brochure
  Arms: Pre-Visit Preparation (PVP) Brochure + QUOCCAS Questionnaire
Diagnostic Test: QUOCCAS Questionnaire — Participants complete the QUOCCAS questionnaire, a structured, self- or caregiver-reported tool designed to identify clinical features, family history, and signs suggestive of cancer predisposition syndromes. Responses are used to classify risk status and are compared against physician-based tools and genetic testing (germline genetic sequencing).
  Other Names: Questionnaire on Congenital Cancer Signs through Self-Assessment
Diagnostic Test: Germline genetic sequencing for Cancer Predisposition Syndromes (CPS) — All participants will provide a saliva or blood sample for germline genetic sequencing. The investigators will perform either whole-exome (WES) or whole-genome sequencing (WGS) and assess for pathogenic/ likely-pathogenic variants in known Cancer Predisposition Genes (CPS).
Diagnostic Test: MIPOGG Assessment — The McGill Interactive Pediatric OncoGenetic Guidelines (MIPOGG) is a clinician-applied digital decision-support tool that uses patient age, tumor type, and clinical features to generate recommendations for referral to genetics. In this study, all participants will undergo MIPOGG assessment performed by the research team through the use of medical records. Results will be compared with those from the QUOCCAS questionnaire to evaluate concordance and potential equivalence in identifying children with cancer predisposition syndromes.

SUMMARY:
This clinical trial tests whether a patient- and caregiver-completed questionnaire (QUOCCAS) can accurately help identify children and adolescents with cancer who may have an underlying cancer predisposition syndrome (CPS). The study will also evaluate whether providing families with an educational brochure before their clinic visit improves their understanding of genetics and their satisfaction with care.

The main questions it aims to answer are:

* Does QUOCCAS identify children at risk for CPS as accurately as physician-based tools and compared to genetic testing?
* Does the Pre-Visit Preparation (PVP) brochure improve caregiver knowledge about genetics?
* Does the PVP brochure improve caregiver satisfaction with the care and information they receive?

Participants will:

* Complete the QUOCCAS questionnaire about family history, clinical features, and cancer signs
* Provide a blood or saliva sample for genetic testing (whole-exome or whole-genome sequencing)
* Randomly receive or not receive the educational Pre-Visit Preparation brochure before completing the questionnaire
* Complete brief surveys on their knowledge and satisfaction

ELIGIBILITY:
Inclusion Criteria:

* The investigators will include newly diagnosed patients who received a cancer diagnosis included in the International Classification of Childhood Cancer version 3 (ICCC3) criteria, treated at participating hospitals

Exclusion Criteria:

* Over 21 years of age

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 205 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the QUOCCAS Questionnaire for Identifying Cancer Predisposition Syndromes (CPS) | Baseline to study completion, up to 36 months
  Accuracy of the QUOCCAS questionnaire in identifying childhood cancer patients at increased risk for a cancer predisposition syndrome, compared to (1) physician standard of care referral, (2) the McGill Interactive Paediatric Oncogenetic Guidelines (MIPOGG), and (3) the gold standard of germline genetic sequencing. Sensitivity is defined as the proportion of CPS cases correctly identified by QUOCCAS; specificity is the proportion of non-CPS cases correctly identified.

SECONDARY OUTCOMES:
Genetic Literacy Score of Caregivers | Baseline to study completion, up to 36 months
  Change in caregiver knowledge and understanding of genetics and cancer predisposition syndromes, measured with a validated genetic literacy questionnaire (Fitzgerald-Butt et al. 2016) and additional CPS-specific items. The genetic literacy score comprises 18 items with each correct item being attributed one point (higher scores from 0-18 indicating higher genetic literacy). The CPS-specific part comprises 10 items with each correctly answered item being attributed one point (higher scores from 0-10 indicating higher genetic literacy). Mean scores of each item will be compared between participants who received the Pre-Visit Preparation (PVP) brochure and those who did not.
Patient and Caregiver Satisfaction with Care and Information | Baseline to study completion, up to 36 months
  Satisfaction measured using the Picker Patient Experience Questionnaire (PPE-15), adapted for the study, focusing on clarity of information, involvement in decision-making, and overall satisfaction with care. Proportions of problematic items (with higher proportions indicating more problematic encounters and negative experience) will be compared between families receiving the PVP brochure and those not receiving it.
Feasibility of Implementing QUOCCAS Questionnaire for Identifying Cancer Predisposition Syndromes and the Pre-Visit Preparation (PVP) Brochure | At study completion, up to 36 months
  Feasibility will be evaluated through the proportion of eligible families who successfully complete the QUOCCAS questionnaire, average time to complete the questionnaire, and provider survey feedback on ease of use and workflow integration.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Waespe, MD PhD, PD, Principal Investigator — University Children's Hospital Bern, Inselspital, Bern, Switzerland
Locations (1):
- Inselspital, Universitäts Kinderklinik (University Children's Hospital) Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Sensitive data on genetic disease of a small patient group which might lead to confidentiality issues. On request, anonymised data can be requested after study completion from the principal investigator.